CLINICAL TRIAL: NCT05566275
Title: Remote Evaluation of Cognitive Function for Older Adults Undergoing Surgery
Brief Title: Remote Cognitive Assessment for Surgical Patients
Acronym: Remote OR
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-28294P; 1RF1AG077557-01 (NIH)
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Mild Cognitive Impairment; Delirium
Keywords: Remote Cognitive Assessment
MeSH Terms: conditions — Cognitive Dysfunction; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a pilot study to evaluate the use of remote cognitive testing to identify patients who may have cognitive vulnerability and may benefit from cognitive care pathways. Participants in this study are asked to complete a smartphone battery of thinking, memory, speech, and motor function tests on their smartphone.

DETAILED DESCRIPTION:
This study is evaluating cognitive function in older adults that are undergoing surgery using remote assessments. Participants complete a battery of neuropsychological assessments prior to their surgery date. The battery includes smartphone adaptions of tests of thinking, memory, speech, and movement. The participant has a one-hour remote visit, where the investigators will conduct a Montreal Cognitive Assessment (MoCA) and have the participant complete the smartphone assessments. After their surgery, participants are evaluated on the delirium rating scale.

ELIGIBILITY:
Inclusion Criteria:

* Spine surgery with a duration greater than or equal to three hours
* Can speak, write, and understand English
* Ability to participate in remote visit

Exclusion Criteria:

* Participating in other cognitive studies
* Having more than one surgery (planned multiday surgery)
* Emergency surgery

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Number of Patients that develop Postoperative Delirium (POD). | Daily after surgery up to discharge from the hospital- an average of days to 2 weeks
  Postoperative Delirium is measured by clinical assessment using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), or the Nursing Delirium Screen Scale (Nu-DESC). A composite delirium score is calculated, and patient is included in the delirium group if either CAM-ICU or NuDESC screenings are positive during the hospital stay. Electronic medical records will also be evaluated for any delirium diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Staffaroni, PhD, Principal Investigator — University of California, San Francisco; Odmara Barreto Chang, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will not make individual participant data available to other researchers.

REFERENCES:
- [Background] Staffaroni AM, Tsoy E, Taylor J, Boxer AL, Possin KL. Digital Cognitive Assessments for Dementia: Digital assessments may enhance the efficiency of evaluations in neurology and other clinics. Pract Neurol (Fort Wash Pa). 2020 Nov-Dec;2020:24-45. No abstract available. PMID 33927583
- [Background] Gaudreau JD, Gagnon P, Harel F, Tremblay A, Roy MA. Fast, systematic, and continuous delirium assessment in hospitalized patients: the nursing delirium screening scale. J Pain Symptom Manage. 2005 Apr;29(4):368-75. doi: 10.1016/j.jpainsymman.2004.07.009. PMID 15857740
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446